CLINICAL TRIAL: NCT00381823
Title: Intervention for Risk Factors in Pregnant Women in Washington, D.C. (DC-HOPE)
Brief Title: Healthy Outcomes of Pregnancy Education
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Children's National Research Institute (Other); Georgetown University (Other); George Washington University (Other); Howard University (Other); RTI International (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: HOPE Study; 3U18HD030445 (NIH); 3U18HD030447 (NIH); 5U18HD031206 (NIH); 3U18HD031919 (NIH); 5U18HD036104 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2006-09-29 (Estimated); Status verified 2006-09

CONDITIONS: Environmental Tobacco Smoke Exposure; Depression; Partner Abuse; Tobacco Smoking
Keywords: Pregnant women; Intervention Studies; African Americans; Infant Mortality; Environmental Tobacco Smoke Pollution; Depression; Partner Abuse; Tobacco Smoke
MeSH Terms: conditions — Depression; Tobacco Smoking; Infant Death | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to determine if an integrated intervention addressing active smoking, environmental tobacco smoke exposure, depression and intimate partner violence, would improve pregnancy outcome among African American women.

DETAILED DESCRIPTION:
This study recruited pregnant, English speaking women from the District of Columbia who were African American or Latina and had one or more of the following risk factors: active smoking, environmental tobacco smoke exposure, depression and intimate partner violence. Women were randomized to receive either an integrated intervention or usual prenatal care. Women randomized to the intervention arm received a cognitive behavioral intervention delivered during the prenatal period in four to eight sessions. Up to two postpartum booster sessions were provided. Sessions were delivered coincident with prenatal care visits. Careful attention was paid to individualizing counseling to provide an integrated approach to each participant's multiple risk factors. The outcomes of interest were primarily behavior change with regard to the risk factors and secondarily to improved birth outcomes, specifically birthweight and gestation.

ELIGIBILITY:
Inclusion Criteria:

* African American or Latina (by self report)
* At least 18 years of age
* English speaking
* Pregnant less than or equal to 28 weeks gestation
* Receiving prenatal care in the District of Columbia
* Had one or more of the following risk factors: active smoking, environmental tobacco smoke exposure, depression and intimate partner violence

Exclusion Criteria:

* Non-minority race (by self report)
* Younger than 18 years of age
* Non-English speaking
* Not pregnant or pregnant greater than 28 weeks gestation
* Receiving prenatal care outside the District of Columbia
* Responded negatively to questions about risk factors
* Suicidal ideation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1750
Dates: Start 2001-07; Study Completion 2004-08

PRIMARY OUTCOMES:
Reduction of risk behaviors:
Active smoking
Environmental Tobacco Smoke Exposure
Depression
Intimate Partner Violence

SECONDARY OUTCOMES:
birth weight
gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Michele Kiely, DrPH, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- Howard University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Hameed M, O'Doherty L, Gilchrist G, Tirado-Munoz J, Taft A, Chondros P, Feder G, Tan M, Hegarty K. Psychological therapies for women who experience intimate partner violence. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013017. doi: 10.1002/14651858.CD013017.pub2. PMID 32608505
- [Derived] Backonja U, Robledo CA, Wallace ME, Flores KF, Kiely M. Reproductive Health Knowledge among African American Women Enrolled in a Clinic-Based Randomized Controlled Trial to Reduce Psychosocial and Behavioral Risk: Project DC-HOPE. Womens Health Issues. 2016 Jul-Aug;26(4):442-51. doi: 10.1016/j.whi.2016.03.005. Epub 2016 Apr 16. PMID 27094910
- [Derived] Kiely M, El-Mohandes AA, Gantz MG, Chowdhury D, Thornberry JS, El-Khorazaty MN. Understanding the association of biomedical, psychosocial and behavioral risks with adverse pregnancy outcomes among African-Americans in Washington, DC. Matern Child Health J. 2011 Dec;15 Suppl 1(Suppl 1):S85-95. doi: 10.1007/s10995-011-0856-z. PMID 21785892
- [Derived] El-Mohandes AA, El-Khorazaty MN, Kiely M, Gantz MG. Smoking cessation and relapse among pregnant African-American smokers in Washington, DC. Matern Child Health J. 2011 Dec;15 Suppl 1(Suppl 1):S96-105. doi: 10.1007/s10995-011-0825-6. PMID 21656058
- [Derived] Molina KM, Kiely M. Understanding depressive symptoms among high-risk, pregnant, African-American women. Womens Health Issues. 2011 Jul-Aug;21(4):293-303. doi: 10.1016/j.whi.2011.01.008. Epub 2011 May 12. PMID 21565525
- [Derived] El-Mohandes AA, Kiely M, Blake SM, Gantz MG, El-Khorazaty MN. An intervention to reduce environmental tobacco smoke exposure improves pregnancy outcomes. Pediatrics. 2010 Apr;125(4):721-8. doi: 10.1542/peds.2009-1809. Epub 2010 Mar 8. PMID 20211945
- [Derived] Kiely M, El-Mohandes AAE, El-Khorazaty MN, Gantz MG. An integrated intervention to reduce intimate partner violence in pregnancy: a randomized controlled trial. Obstet Gynecol. 2010 Feb;115(2 Pt 1):273-283. doi: 10.1097/AOG.0b013e3181cbd482. PMID 20093899
- [Derived] El-Mohandes AA, Kiely M, Gantz MG, Blake SM, El-Khorazaty MN. Prediction of birth weight by cotinine levels during pregnancy in a population of black smokers. Pediatrics. 2009 Oct;124(4):e671-80. doi: 10.1542/peds.2008-3784. Epub 2009 Sep 28. PMID 19786427